CLINICAL TRIAL: NCT03002779
Title: A Phase 1, Open Label Study to Characterize the Absorption, Metabolism and Excretion of 14C-JNJ-53718678 After a Single Dose in Healthy Adult Male Subjects
Brief Title: A Study to Characterize the Absorption, Metabolism, and Excretion of 14C-JNJ-53718678 After a Single Oral Dose in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108210; 53718678RSV1008 (Other: Janssen Research & Development, LLC); 2016-002664-14 (EudraCT Number)
Record Dates: First submitted 2016-11-30; First posted 2016-12-26 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-53718678

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JNJ-53718678 (Experimental)
  Interventions: Drug: JNJ-53718678

INTERVENTIONS:
Drug: JNJ-53718678 — Participants will receive a single 500 milligram (mg) dose of 14C-JNJ-53718678 as an oral liquid solution containing 14C-labeled and unlabeled JNJ-53718678 corresponding to a radioactivity dose.

SUMMARY:
The purpose of the study is to determine the routes of excretion for JNJ-53718678 and its metabolites, to explore the metabolic pathways of JNJ-53718678, and to determine the chemical structure of predominant metabolites in healthy adult male participants after a single oral dose of 500 milligram (mg) 14C-JNJ-53718678.

ELIGIBILITY:
Inclusion Criteria:

* A male participant: a) Must be sexually abstinent (defined as refraining from sexual intercourse from Day 1 (day of dosing) until 90 days after study drug administration), OR b) Who is sexually active (either heterosexual, including with a pregnant woman, or homosexual) must agree to use a barrier method of contraception (eg, condom) from Day 1 (day of dosing) until 90 days after study drug administration, AND c) Who is sexually active with a woman of childbearing potential must agree to use a barrier method of contraception (eg, condom) from Day 1 (day of dosing) until 90 days after study drug administration, in conjunction with this female partner using a highly effective contraceptive (such as implantable progestogen-only hormone contraception associated with inhibition of ovulation; intrauterine device; intrauterine hormone-releasing system, combined [estrogen- and progestogen- containing] hormonal contraception associated with inhibition of ovulation: oral, intravaginal, or transdermal; progestogen-only hormone contraception associated with inhibition of ovulation: oral or injectable) d) Must agree not to donate sperm from Day 1 (day of dosing) until 90 days after study drug administration
* Participant must have a body mass index (BMI; weight in kg divided by the square of height in meters) of 18.0 to 30.0 kilogram per square meter (kg/m^2)
* Participant must have a blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic
* Participant must have a normal 12-lead electrocardiogram (ECG) (based on the mean value of triplicate ECG parameters), consistent with normal cardiac conduction and function at screening, including: a) normal sinus rhythm (heart rate between 45 and 90 beats per minute (bpm), extremes included); b)mean QT interval corrected for heart rate according to Fridericia formula (QTcF) interval lesser than or equal to (<=)450 millisecond (ms); c) mean QRS interval of <110 ms; d) mean PR interval <200 ms; e) morphology consistent with healthy cardiac conduction and function
* Participants must be healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination (including height and body weight measurement and skin examination), medical history, vital signs (systolic and diastolic blood pressure, pulse rate, orthostatic blood pressure changes, respiratory rate, and body temperature), creatinine clearance (below 60 milliliter per minute (mL/min) at screening using Cockroft-Gault equation), and the results of blood biochemistry, blood coagulation, and hematology tests, and a urinalysis performed at screening, on Day -1, or predose on Day 1, whichever is applicable. If there are abnormalities, with the exception of those described in the in- and exclusion criteria, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator

Exclusion Criteria:

* Participants with a removed gallbladder, or with a history of upper gastrointestinal (stomach, duodenum) surgery, or with a recent (less than 3 months prior to screening) episode of gallbladder stones
* Participants with a history of heart arrhythmias (extrasystoles, tachycardia at rest) or history of risk factors for Torsade de Pointes syndrome (example, hypokalemia, family history of long QT syndrome)
* Participant has intolerance to xylocaine, lactose, or midazolam
* Participant has a history of hepatitis A antibody immunoglobulin M (IgM), hepatitis B virus surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for hepatitis A antibody IgM, HBsAg or anti HCV at screening
* Participant has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Mass Balance of JNJ-53718678 in Healthy Adult Male Participants. | Up to Day 10
  Total mass balance calculated by D(dose) urine, total (percent [%]) + D feces, total (%) + D duodenal, total (%) where D urine, total is the total percentage of the dose excreted into urine, calculated as 100 * (Ae total [total amount excreted into urine, calculated by adding the amounts of the individual intervals together] /Dose); D feces,total is the total percentage of the dose excreted into feces, calculated as 100 * (Ae total [total amount excreted into feces, calculated by adding the amounts of the individual stools together]/Dose) and D duodenal, total is defined as total percentage of the dose collected in all duodenal samples collectively, calculated as % of dose.
Metabolic profiles of JNJ-53718678 in plasma, duodenal fluid, urine, and feces samples with radio high-performance liquid chromatography analysis | Up to Day 6
  Metabolite profiling will be performed with radio high-performance liquid chromatography.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Throughout the study duration (up to 24 days)
  Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences Onderzoekscentrum Groningen, locatie Martini, Groningen, Netherlands